CLINICAL TRIAL: NCT06470620
Title: The Relationship Between Pelvic Floor Muscle Function and Hip Pain Among Women
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PHD, Prof., University of Haifa
Other Study IDs: 122/24
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Incontinence Stress; Incontinence; Hip Pain Chronic
Keywords: pelvic floor; women health; ultrasound; incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- research group: women with hip-related pain
  Interventions: Diagnostic Test: pelvic floor muscle assessment
- control group: healthy women without hip pain
  Interventions: Diagnostic Test: pelvic floor muscle assessment

INTERVENTIONS:
Diagnostic Test: pelvic floor muscle assessment — no intervention will be performed - several diagnostic assessments tools
  Other Names: abdominal ultrasound

SUMMARY:
This study examines the relationship between pelvic floor muscle (PFM) function and self-perception of PFM contraction with hip pain, their severity, and hip muscle strength.

In addition, it will examines the association between PFM function, and anxiety.

DETAILED DESCRIPTION:
This cross-sectional study will include women with symptoms of hip-related pain persisting > three months(research group), and women without hip pain (control group). A single session will include various assessments as follows: abdominal ultrasound examination to evaluate PFM function and endurance, in addition, each participant will evaluate her ability to perform correct contraction of PFM, hand-held dynamometer testing for hip rotator muscle strength, the International Consultation on Incontinence Questionnaire (ICIQ) for evaluating symptoms and impact of urinary incontinence, the International Hip Outcome Tool 12 for assessing hip function and pain, the Hospital Anxiety & Depression Scale (HADS), and a functional performance task involving the hip muscles - a single-leg squat.

ELIGIBILITY:
Inclusion Criteria for Research Group:

* complaints of hip related pain,
* Visual Analog Scale (VAS) >3 for three months,
* with one or more of the symptoms relevant to the syndrome - (1) hip or groin pain produced by a certain movement or position, stiffness and limitation of movement or clicks from the hip joint, (2) examination A positive FADIR performed by the researcher before conducting the study

Exclusion criteria:

* the presence of additional diagnoses of the slipped capital femoral epiphysis,
* Perthes disease,
* avascular necrosis, and osteoarthritis-Calve-Legg,
* neurological or Metabolism,
* surgery/fracture in the hip joint of which the woman complains,
* pregnancy or childbirth in the last year,
* Treatment of the pelvic floor in the last year.

control group - health women without any pain or symptoms in the spine and lower extremities

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the study examine pelvic floor muscle function among women
Study Population: women with and without hip related pain
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire | baseline
  evaluating the frequency, severity and impact on quality of life of urinary incontinence. The score ranges from 0-21, with a higher score indicating greater severity
pelvic floor muscle function assessed as correct movement of the urinary bladder | baseline
  upward or downward displacement of urinary bladder will be measured via diagnostic ultrasound. Upward movement is considered the correct direction describing good function of pelvic floor muscles
urinary bladder displacement in millimeters | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool
pelvic floor muscles endurance of contraction in seconds | baseline
  The participant is instructed to contract pelvic floor muscle and hold the contraction as long as possible. bladder status on ultrasound is assessed. When the bladder starts to move downward from its position the examination ends. (measured in sec).

SECONDARY OUTCOMES:
muscle strength | baseline
  hip muscle abduction sill be measure via hand held dynamometer
hip function assessment | baseline
  International Hip Outcome Tool 12 questionnaire. range 0-100, with a high score indicates a high quality of life
self-reporting of fear and anxiety of hip pain regarding quality of life | baseline
  Hospital Anxiety & Depression Scale
hip range of motion | baseline
  range of motion will be assessed with goniometer
function assesment | baseline
  single leg squat

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Haifa District, Israel

IPD SHARING:
Plan to Share IPD: Yes
following study completion, a paper will be submitted to international professional journal
Supporting Information: Study Protocol, CSR
Time Frame: 6 months following end of study

REFERENCES:
- [Result] Dar G, Saban TS. The Perception of Pelvic Floor Muscle Function amongst Exercising Women Who Are Repeatedly Instructed to Contract Their Pelvic Floor Muscles. Healthcare (Basel). 2022 Sep 14;10(9):1768. doi: 10.3390/healthcare10091768. PMID 36141380